CLINICAL TRIAL: NCT07105462
Title: Application of Intelligent Visual Training in the Sports Industry: The Effects of Rotational Prisms on Badminton Players' Ocular Vergence Training and Enhancement of Shot Accuracy
Brief Title: The Effects of Rotational Prisms on Badminton Players' Ocular Vergence Training and Enhancement of Shot Accuracy
Acronym: ADRRPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRREC-114-011
Record Dates: First submitted 2025-07-16; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Eye Movements; Visual Perception; Psychomotor Performance; Sports

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Vergence Training with ADRRPs (Experimental): Participants assigned to this arm will receive vergence training using Automatic Dual Rotational Risley Prisms (ADRRPs), a computerized visual device designed to induce alternating base-out and base-in prism stimulation. The prisms rotate automatically to simulate dynamic convergence and divergence demands, cycling between 0 to 30 prism diopters base-out over 5 seconds and 30 base-out to 10 base-in over 3 seconds. Each participant will undergo 8 training sessions over 4 weeks (twice weekly), with each session lasting 15 minutes. During training, participants view standardized video targets positioned at a 40 cm working distance while instructed to maintain clear and single binocular vision. The intervention aims to engage and strengthen vergence eye movements critical for visual performance in dynamic sports environments.
  Interventions: Device: Arm 1 - Experimental Group Intervention Name: ADRRPs Vergence Training Intervention Description: Participants wore an Automatic Dual Rotational Risley Prism (ADRRPs) headset to perform vergence eye
- Arm 2: Sham Training with Plano Lenses (Sham Comparator): Participants assigned to this arm will undergo sham vergence training using the same Automatic Dual Rotational Risley Prisms (ADRRPs) headset, but fitted with non-refractive plano lenses and with no prism rotation. The training schedule and environment are identical to the intervention arm: 8 sessions over 4 weeks (twice weekly), with each session lasting 15 minutes. Visual targets are presented at a 40 cm viewing distance using the same video stimuli. This sham training condition is designed to control for potential placebo effects and to isolate the specific influence of dynamic prism-induced vergence stimulation used in the experimental arm.
  Interventions: Device: 1. Experimental Group Intervention Name: ADRRPs-Based Vergence Training; 2. Control Group Intervention Name: Sham Training with Plano Lenses.

INTERVENTIONS:
Device: Arm 1 - Experimental Group Intervention Name: ADRRPs Vergence Training Intervention Description: Participants wore an Automatic Dual Rotational Risley Prism (ADRRPs) headset to perform vergence eye — ADRRPs Vergence Training
  Intervention Description:
  Participants wore an ADRRPs headset that applied alternating base-in and base-out prism power to stimulate vergence eye movements. Prism levels were customized based on each participant's fusional vergence. Training was performed twice weekly for 15 minutes over four weeks while viewing a near video target.
  Sham Visual Training with Plano Lenses
  Intervention Description:
  Participants wore an identical ADRRPs headset fitted with plano lenses that produced no prism effect. The procedure and schedule matched the experimental group but provided no vergence stimulation, serving as a sham control.
  Arms: Arm 1: Vergence Training with ADRRPs
Device: 1. Experimental Group Intervention Name: ADRRPs-Based Vergence Training; 2. Control Group Intervention Name: Sham Training with Plano Lenses. — ADRRPs-Based Vergence Training This intervention used the Automatic Dual Rotational Risley Prisms (ADRRPs) system to deliver alternating base-in and base-out prism stimulation for vergence training. Prism levels were customized based on each participant's fusional vergence. Training was conducted twice per week for four weeks, 15 minutes per session, while participants viewed a near video target. This protocol provides automated and symmetric vergence demand, distinguishing it from conventional near-point or static prism exercises.
  Sham Training with Plano Lenses Participants used the same ADRRPs headset as the experimental group but with plano lenses that produced no prism effect. The training schedule and visual tasks matched the experimental condition, but no vergence stimulus was applied. This design enabled participant masking while providing no active optical stimulation, serving as a sham comparator distinct from both active training and no-treatment controls.
  Arms: Arm 2: Sham Training with Plano Lenses

SUMMARY:
This randomized controlled trial is designed to investigate whether a novel visual training system can improve eye coordination, reaction time, and hitting accuracy in competitive badminton players. The training utilizes a device called the Automatic Dual Rotational Risley Prisms (ADRRPs), which presents alternating base-in and base-out prism demands to stimulate vergence eye movements. This type of training aims to enhance the eyes' ability to converge and diverge quickly and accurately-a function that is important for visual clarity and motor performance during fast-paced sports.

A total of 26 collegiate badminton athletes aged 18 to 25 years will be recruited from two universities in Taiwan. Participants will be randomly assigned to one of two groups: a visual training group using the active ADRRPs system, and a control group using a sham version of the same device containing plano lenses (with no prism effect). Training will be delivered twice per week for four weeks, with each session lasting 15 minutes. During each session, participants will view a video while the device applies alternating prism stimulation based on each individual's pre-measured fusional vergence capacity.

Outcome measures will be assessed at baseline and after the four-week training period. These include vergence facility (cycles per minute), accommodative facility (flipper test), near point of convergence, and positive fusional vergence at near. Reaction time will be measured using a light-based agility task with BlazePod sensors, and hitting performance will be evaluated using a shuttlecock launcher that delivers randomized targets to various court zones.

All participants will be monitored for any adverse events, and any symptoms such as diplopia, dizziness, or discomfort will be documented. Data will be analyzed as described in the Statistical Analysis Plan.

DETAILED DESCRIPTION:
This randomized controlled trial explores the application of vergence eye movement training in enhancing visuomotor performance in competitive badminton athletes. The intervention utilizes a device known as the Automatic Dual Rotational Risley Prisms (ADRRPs), which delivers alternating base-out and base-in prism stimulation in an automated manner to engage binocular vergence mechanisms.

The study targets young adult badminton players with at least two years of consistent training. Participants are randomly allocated to either an experimental group, which receives active prism training using the ADRRPs, or a control group using an identical headset without prism rotation. Both groups undergo training sessions twice a week for four weeks, with each session lasting 15 minutes. Visual stimuli are standardized across groups and delivered at a fixed near working distance of 40 cm.

The prism rotation parameters are set to simulate dynamic vergence demands based on pre-measured individual capabilities. This approach aims to create a structured vergence load while minimizing visual discomfort. The control condition serves to control for placebo and attentional effects.

Outcome measures are selected to assess both oculomotor and performance domains. These include vergence facility, accommodative facility, near point of convergence, and positive fusional vergence-all measured using standardized optometric tools. Reaction time is assessed via a BlazePod light stimulus test, and hitting accuracy is evaluated through a shuttlecock launcher delivering randomized trajectories to simulate game-like performance.

The trial design incorporates single-blinding and concealed allocation procedures. Data analysis will follow a pre-specified statistical analysis plan, and participants will be closely monitored for any adverse symptoms during the course of the intervention. Ethics approval has been obtained from the relevant institutional review board.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years
* Minimum of 2 years of consistent badminton training
* Best-corrected visual acuity of 20/25 or better in both eyes (distance and near)
* No history of ocular pathology
* Willingness to comply with all study procedures and follow-up

Exclusion Criteria:

* Presence of constant strabismus or binocular vision anomaly
* History of ocular trauma, strabismus surgery, or refractive surgery
* Neurological or systemic conditions affecting vision
* Ongoing medication that may influence ocular motor function

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Reaction Time Measured by BlazePod Test | Baseline and Week 4 (post-intervention)
  * Time in seconds required to complete 10 light-response trials using BlazePod; lower values indicate better performance.
  * Unit of Measure: seconds

SECONDARY OUTCOMES:
Vergence Facility in Cycles per Minute (cpm) | Baseline and Week 4
  * Measured using 12 BO/3 BI prism flippers at 40 cm with a 20/32 target; higher values indicate better vergence flexibility.
  * Unit of Measure: cycles per minute
Accommodative Facility in Cycles per Minute (cpm) | Baseline and Week 4
  * Measured binocularly with ±2.00 D flippers at 40 cm.
  * Unit of Measure: cycles per minute
Near Point of Convergence Distance | Baseline and Week 4
  * Break point measured using RAF rule.
  * Unit of Measure: centimeters
Positive Fusional Vergence Break and Recovery Points | Baseline and Week 4
  * Measured using prism bars at 40 cm. Report break and recovery values.
  * Unit of Measure: prism diopters
Number of Successful Shuttlecock Hits | Baseline and Week 4
  * Number of accurate hits out of 16 randomized shuttle launches.
  * Unit of Measure: count (number)

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Yu Huang, Ph.D., Study Chair — College of Health Sciences, Central Taiwan University of Science and Technology
Locations (1):
- Central Taiwan University of Science and Technology, Taichung, Taiwan